CLINICAL TRIAL: NCT05643274
Title: Use of Long Read Genome Sequencing in Patients Suffering From Neurodevelopmental Troubles
Acronym: HiFi-NDD
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Rennes University Hospital (Other); University Hospital, Angers (Other Government); University Hospital, Brest (Other); University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RC22_0373
Record Dates: First submitted 2022-11-22; First posted 2022-12-08 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Genetic Disease; Neurologic Disorder; Developmental Delay Disorder; Growth Disorders
Keywords: long read sequencing; rare genetic diseases; neurodevelopmental diseases; diagnostic
MeSH Terms: conditions — Genetic Diseases, Inborn; Nervous System Diseases; Developmental Disabilities; Growth Disorders; Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Patients with neurodevelopmental disease and their both parents

SUMMARY:
Patients with neurodevelopmental diseases and their families need to identify the genetic cause of the disease to allow for recognition of the disability, genetic counseling, and possible hope for participation in therapeutic research studies. Access to high-throughput genomic exome or genome analysis allows the identification of a genetic cause for approximately half of the patients. However, families with no result or with a variant of unknown significance after these tests may find themselves in a new diagnostic impasse.

The high-throughput sequencing used today generates sequences of the order of 100 base pairs (so-called "short read" sequencing). This allows an analysis of about 90% of the genome. However, many regions are not accessible in regions of interest for the genetic diagnosis of rare diseases. Long fragment sequencing generates sequences that are about 20 times larger and its use has recently made it possible to sequence the human genome almost completely (https://www.science.org/doi/10.1126/science.abj6987). The main contribution lies in the analysis of complex regions of the genome such as segmental duplications or centromeric regions. It is likely that this technology increases the sensitivity of detection of genetic variants in patients with genetic diseases. Its contribution should be studied in patients for whom no genetic cause has been identified by classical techniques.

This study aim to investigate the contribution of long fragment genome sequencing.

DETAILED DESCRIPTION:
Ten families with a child suffering from a neurodevelopmental disease will be recruited by geneticists being part of the CLAD-Ouest. An EDTA blood sample will be taken from the patient and their parents (trio analysis). The blood samples will then be used to extract nucleic acids (DNA).

The blood samples will be sent and centralized to the genetics laboratory of the Nantes University Hospital. The DNA will be extracted and anonymized.

The files generated after DNA sequencing will have as an identification key the anonymization number provided at the time of inclusion of the individual in the study. The raw data and VCF files will be uploaded to the BIRD computing cluster in Nantes, where they will be stored for the duration of the study (2 years). The different university hospitals will then be able to retrieve the data and analyze the variants identified in the patients recruited by their center. A centralized analysis to annotate, filter and interpret the variants will be performed by a group of bioinformaticians and biologists from HUGO (University Hospital from the Grand Ouest). Long-term archiving of the data will be performed at the Nantes University Hospital.

ELIGIBILITY:
Inclusion Criteria for patients:

* Patient (child or adult) presenting neurodevelopmental troubles strongly suspected to suffer from a rare genetic disease (familial or very severe).
* Negative outcome for short read sequencing of the trio (child and parents).
* Informed consent to the study by the patient (if applicable) or their legal representatives if under-aged or under guardianship.
* Patients benefiting from the social security (French health care system).

Inclusion criteria for Parents :

* Possible recruitment of both parents matching the inclusion criteria.
* Informed consent form signed for their own participation.
* Parents benefiting from the social security (French health care system).

Exclusion Criteria for patients:

* Genetic predisposition already identified explaining the disease.
* Paients for which the WGS for the trio has not been performed.
* Patients having withdrawn their consent.

Exclusion Criteria fo Parents :

* Pregnant or lactating woman.
* Parents under guardianship or curatorship.
* Parents also presenting a neurodevelopmental deficiency.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient with neurodevelopmental diseases and their both parents
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Use of long read sequencing in patients suffering from a neurodevelopmental disease without pathogenic or probably pathogenic variation identified by short read sequencing | through study completion, an average of 2 years
  Identification of a genetic diagnosis : detection of one or several variant(s) - nucleotidic, change in copy number, structural variants- of class 4 or 5 (probably pathogenic or pathogenic), explaining the genetic origin of the neurodevelopmental pathology

SECONDARY OUTCOMES:
Analysis of the implementation of the long read sequencing of trios (patients and parents) | through study completion, an average of 2 years
  Measurement of the failing rate of long read sequencing, turn around time between sequencing and results available to clinical team

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane BEZIEAU, MD, Principal Investigator — Nantes University Hospital
Locations (5):
- France (5):
  - Brest University Hospital, Brest, Finistère
  - Rennes University Hospital, Rennes, Ille-et-Vilaine
  - Tours University Hospital, Tours, Indre-et-Loire
  - Nantes University Hospital, Nantes, Loire-Atlantique
  - Angers University Hospital, Angers, Maine-et-Loire

IPD SHARING:
Plan to Share IPD: Undecided